CLINICAL TRIAL: NCT02618213
Title: Comparison of High Flow Oxygenation Therapy and CPAP in Children With Bronchiolitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Signe Voss Vahlkvist, MD PhD, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20150007
Record Dates: First submitted 2015-11-25; First posted 2015-12-01 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Respiratory Syncytial Virus Bronchiolitis
Keywords: Continuous Positive Airway Pressure; High Flow Oxygenation therapy; Bronchiolitis; Children
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continous Positive Airway Pressure (Active Comparator): CPAP is administered through a binasal tube fitted with a Benveniste gas jet administered with humified airflow. Start flow is 12-14 l/min and can be changed to maximum 15 or minimum 12 l/min. Oxygen can be supplied as needed to keep SpO2 (peripheral capillary Oxygen saturation) within acceptable limits.
  Interventions: Device: Continous Positive Airway Pressure
- High Flow Oxygenation Therapy (Active Comparator): HFOT is administered by optiflow Junior ( Fisher&Paykal Healthcare® Auckland, New Zealand) Start flow 12-14 l/min. Oxygen can be supplied as needed to keep Sp02 within acceptable limits
  Interventions: Device: Optiflow Junior

INTERVENTIONS:
Device: Optiflow Junior — Humified air are dispensed through the system. Airflow, FiO2 (Fraction of inspired oxygen) , SpO2 (peripheral capillary Oxygen saturation) and respiratory rate are noted each hour. Progression of condition might lead to change of system og mechanical ventilation. poor tolerance might lead to change of system
  Other Names: High Flow Oxygenation Therapy; HFOT
  Arms: High Flow Oxygenation Therapy
Device: Continous Positive Airway Pressure — Humified air are dispensed throug the system. Airflow, FiO2, SpO2 and respiratory rate are noted each hour. Progression of condition might lead to change of system or mechanical ventilation. Poor tolerance might lead to change of system.
  Other Names: CPAP
  Arms: Continous Positive Airway Pressure

SUMMARY:
Bronchiolitis in infants and young children often requires respiraty support. In Denmark Continous Positive Airway Pressure ( CPAP) are routinely used in children with moderate-severe bronchiolitis. The aim of the study is to compare CPAP and High Flow Oxygenation Therapy (HFOT) as tools of respiratory support in infants and young children with bronchiolitis.

Infants and young children with moderate-severe bronchiolitis and are randomized to either CPAP or HFOT.

ELIGIBILITY:
Inclusion Criteria:

* infants and children with moderate respiratoric syncytial virus bronchiolitis or other viral bronchiolitis and need of respiratory support. ( clinical decision)

Exclusion Criteria:

* severe bronchiolitis with P C02 > 9, decreased consciusness and risk for early progression to intensive therapy.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
respiration rate | after 6 12 18 24 and 48 hour of intervention
  change in respiration rate ( RR) from preintervention value
PCo2 | after 6 12 24 and 48 hours of intervention
  Change in PCo2 (partial pressure of carbon dioxide)from pre intervention value
Modified asthma score (MWAS) | Once daily as long as intervention precedes ( 1-14 days)
  Change in MWAS from pre intervention value

SECONDARY OUTCOMES:
treatment length | from beginning of intervention to discontinuation (1-14 days)
  duration of need of intervention ( hours)
Hspitalization | from hospitalization to release (1-21 days)
  duration of hospitalisation ( days)
Intervention failure. | from beginning of intervention to discontinuation.(1-14 days)
  numbers of intervention failure defined as change of intervention or progression to need for intensive care/ mechanical ventilation.
patient acceptance of intervention | daily VAS score (0-5) from beginning of intervention to discontinuation (1-14 days)
  VAS score of tolerance with intervention. 0 = worst possible acceptance 5 = fully acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Signe VAhlkvist, MD PhD, Principal Investigator — Pediatric Award, Hospital of South West Denmark
Locations (2):
- Denmark (2):
  - Hospital Lillebaelt, Kolding
  - Signe Vahlkvist, Kolding